CLINICAL TRIAL: NCT06441344
Title: First-line Etoposide Combined With Platinum-based Chemotherapy Followed by Toripalimab Plus Anlotinib for the Maintenance of Extensive Stage Small Cell Carcinoma - A Randomized, Controlled, Multicenter Phase III Clinical Study
Brief Title: Toripalimab Plus Anlotinib for the Maintenance of Extensive Stage Small Cell
Acronym: SCLC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Dongqing Lv, MD, Chief medical officer, Taizhou Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCLC-maintaine
Record Dates: First submitted 2024-03-19; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: SCLC; Maintenance Treatment
Keywords: ES-SCLC; Maintenance Treatment; Toripalimab; Anlotinib
MeSH Terms: interventions — toripalimab; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- platinum+etoposide → toripalimab plus anlotinib (Experimental): The experimental group was given etoposide (100 mg/m2) d1-3+carboplatin (AUC 5 d1)/cisplatin (25 mg/m2)d1-3 Chemotherapy regimen, for patients who have received 4-6 cycles chemotherapy sessions (including PR, CR, SD), they will enter the maintenance treatment phase and receive an oral dose of 12 mg of anlotinib (d1-14) combined with intravenous infusion of toripalimab 240mg for maintenance treatment until progress or intolerable adverse reactions occur or died for other illnesses
  Interventions: Drug: Toripalimab plus Anlotinib
- platinum+etoposide+ toripalimab → toripalimab (Active Comparator): The control group was given etoposide (100 mg/m2) d1-3+carboplatin (AUC 5) d1/cisplatin (25mg/m2)+and toripalimab (240 mg) ,for patients who have received 4-6 cycles chemotherapy sessions (including PR, CR, SD), they will enter the maintenance treatment phase and receive maintenance treatment with toripalimab 240 mg d1 until progress or intolerable adverse reactions occur or died for other illnesses
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab plus Anlotinib — For patients who did not progress after standard chemotherapy, toripalimab plus anlotinib maintenance therapy was used
  Arms: platinum+etoposide → toripalimab plus anlotinib
Drug: Toripalimab — For patients who did not progress after standard chemotherapy+toripalimab, toripalimab maintenance therapy was used
  Arms: platinum+etoposide+ toripalimab → toripalimab

SUMMARY:
This is a randomized, open, multicenter Phase III clinical study. A total of 136 participants are planned to be enrolled and randomly assigned to either the experimental group (platinum+etoposide → toripalimab plus anlotinib) or the control group (platinum+etoposide+ toripalimab → toripalimab) in a 1:1 ratio. The primary efficacy measures include PFS, while secondary endpoints include OS, DOR, ORR, DCR, progression free survival at 6 and 12 months, overall survival at 12 and 18 months, health-related quality of life (FACT-L), safety, etc. And in the III clinical study, tissue samples were collected before treatment, and tumor tissue and blood samples were taken from some patients after 3 cycles of maintenance treatment and treatment progression for single-cell sequencing and transcriptome sequencing to verify the underlying mechanism research

DETAILED DESCRIPTION:
This study plans to enroll 136 subjects and randomly allocate them in a 1:1 ratio to the experimental group (platinum+etoposide → toripalimab plus anlotinib) and the control group (platinum+etoposide+ toripalimab → toripalimab). The experimental group was given etoposide (100 mg/m2) d1-3+carboplatin (AUC 5 d1)/cisplatin (25 mg/m2 D1-3) chemotherapy regimen, for patients who have received 4-6 cycles chemotherapy sessions (including PR, CR, SD), they will enter the maintenance treatment phase and receive an oral dose of 12 mg of anlotinib ( on days 1-14) combined with 240 mg toripalimab for maintenance treatment; The control group was given etoposide (100 mg/m2) d1-3+carboplatin (AUC 5) d1/cisplatin (25mg/m2) d1+toripalimab 240 mg d1 (including PR, CR, SD) who have been treated 4-6 cycles will enter the maintenance treatment period, and receive maintenance treatment with toripalimab 240 mg d1 . The above treatment regimen lasts for 21 days per cycle until disease progression or Intolerable adverse reactions occur or researchers believe that patients are not suitable for continued medication. After the subject terminates or withdraws from this study, the researcher may adopt reasonable follow-up treatment based on the subject's condition. All patients will be followed up until death or the deadline for data collection. Collect pathological tissue samples before treatment for genetic testing. Before using maintenance therapy medication, after 1 cycle of maintenance therapy and during progression, after 3 cycles of treatment, some patients are selected for puncture biopsy sampling after treatment progression Perform sequencing and biomarker inspection. Follow up on PFS, OS, ORR, DCR, adverse reactions, etc. in two groups of patients. Before maintenance therapy, researchers are allowed to perform local radiotherapy based on the patient's actual situation, such as cranial radiotherapy, bone metastasis radiotherapy, etc., but radiotherapy for the target lesion is not allowed. However, additional treatments related to tumors, including traditional Chinese medicine and radiation therapy, are not allowed during the maintenance treatment process. The primary endpoints of this study were objective progression free survival (PFS) and overall survival (OS) evaluated according to the RECIST v1.1 criteria, while secondary endpoints were duration of response (DOR), overall objective response rate (ORR), disease control rate (DCR)and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 and<80 years old.
* The ECOG score is 0-1 points (including 0 and 1 points), and the expected survival period is not less than 3 months.
* Confirmed as small cell lung cancer (SCLC) by histopathology or cytology and diagnosed as extensive after systemic evaluation.
* I have not received first-line treatment for ES-SCLC systemic chemotherapy or immune checkpoint inhibitors in the past.
* Limited stage SCLC progresses to extensive stage SCLC after receiving previous radiotherapy and chemotherapy aimed at cure,at least 6 months of no treatment period is required after the last radiotherapy and/or chemotherapy treatment.
* Patients with previous active brain metastases have stabilized after treatment and do not require immediate or planned brain intervention during the study period Transfer for local treatment.
* According to the criteria for evaluating the efficacy of solid tumors (RECIST v1.1), enrolled patients should have at least one tumor throughout their body The tumor lesion can meet the following requirements: it has not undergone local treatment such as radiotherapy in the past and is at baseline Can be accurately measured, with a baseline maximum diameter of ≥ 10mm (if it is a lymph node, a minimum diameter of ≥ 15mm is required).

Lesions that have previously received local treatment (radiotherapy or other treatments), if the treatment is completed for at least 6 months If disease progression occurs later, the lesion in the area that has undergone local treatment can be considered a measurable lesion.

* Patients should have sufficient bone marrow reserve function and no liver, kidney, or coagulation dysfunction, and laboratory tests should be conducted
* The value must meet the following conditions:

  1. Absolute neutrophil count ≥ 1.5 × 109/L, and white blood cell count ≥ 3 × 109/L;
  2. Platelet count ≥ 100 × 109/L;
  3. Hemoglobin ≥ 90g/L;
  4. Serum creatinine (Cr) ≤ 1.5 x Upper limit of normal (ULN) or creatinine clearance rate (CrCl) ≥ 50ml/min (for patients with serum creatinine>1.5 x ULN);
  5. If there is no confirmed liver metastasis, AST and ALT ≤ 2.5 × ULN; If there is confirmed liver metastasis, AST,ALT ≤ 5 × ULN;
  6. If there is no confirmed liver metastasis, total bilirubin ≤ 1.5 × ULN; If there is confirmed liver metastasis or patients with syndrome (high indirect bilirubinemia), total bilirubin ≤ 3 x ULN;
  7. If there is no confirmed liver metastasis, alkaline phosphatase (ALP) ≤ 2.5 x ULN or ≤ 5 x ULN (bone metastasis)
  8. Albumin (ALB)>30g/dl;
  9. 24-hour urine protein quantification<1g (if urine protein ≥ 2+, additional 24-hour urine protein testing is required)
  10. Serum lipase or amylase ≤ 1.5 x ULN or>1.5 x ULN (clinical or imaging diagnosis of pancreas)
  11. International standardized ratio (INR) ≤ 1.5, and activated partial prothrombin time (APTT)≤ 1.5 x ULN.
* Female subjects with reproductive ability have a negative blood pregnancy result within 7 days before starting the study treatment, and are willing to From the time of signing the informed consent form until the end of the last medication use, abstain from sexual activity or take medication for a period of 6 months medically recognized and efficient contraceptive measures (such as intrauterine devices, condoms, etc.), but the use of hormones is prohibited Using similar drugs for contraception; Male subjects are willing to take informed consent from the time of signing until the end of the last medication use Within the next 6 months, abstain from sexual activity or use medically recognized and effective contraceptive measures (such as condoms),and during this period, no sperm will be donated;.
* The subjects are able to understand and voluntarily sign a written informed consent form (the informed consent form must be completed before conducting the study) Sign before any program specified in the plan.
* Be able to voluntarily complete the research procedures and follow-up examinations according to the requirements of the research protocol.

Exclusion Criteria:

* Mixed small cell lung cancer diagnosed by histology or cytology;
* A history of severe allergic diseases, severe drug (including unmarketed investigational drugs) allergies, or known adverse reactions to this medication Allergy to any component of the investigational drug: presence of etoposide, platinum based drugs (carboplatin/cisplatin), or anlotinib.Individuals who are contraindicated to the use of anlotide or Toripalimab;
* Previously received treatment with immune checkpoint agonists (such as CD137 agonists) or immune checkpoint inhibitors.Preparation therapy (such as single/dual antibodies against CTLA-4, PD-1, PD-L1, LAG3, etc.) or anti VEGF targeted drugs;
* Previously received curative radiotherapy (excluding those who met the inclusion criteria of 5), or before receiving study treatment.Has undergone extensive palliative radiotherapy within 4 weeks, or plans to undergo chest radiotherapy during the study period
* Need or plan to undergo elective surgical treatment during the trial period;
* Received the following treatments or medications before starting the research treatment:

  1. Received important organ surgery (excluding puncture) within 28 days before starting the study and treatment Inspection;
  2. Received attenuated live vaccine within 28 days prior to starting treatment;
  3. Have used intravenous broad-spectrum antibiotics for at least 7 days within 14 days before starting the study treatment;
  4. Starting the study on systemic corticosteroids (prednisone>10) received within 14 days prior to treatment Mg/day or equivalent dose of similar drugs or other immunosuppressive treatments; Except for the following situations External: Treatment with local, ocular, intra-articular, intranasal, and inhaled corticosteroids; short Regular use of glucocorticoids for preventive treatment (such as preventing contrast agent allergies);
  5. Received palliative radiotherapy for bone metastases within 14 days prior to starting the study treatment;
* Currently, there is spinal cord compression or superior vena cava syndrome;
* Currently, there are clear cases of interstitial lung disease or non infectious pneumonia, except for those caused by local radiotherapy;
* There are brain metastases in the midbrain, pons, medulla oblongata, spinal cord, meninges, and meninges, or symptomatic large brain metastases Brain or cerebellar metastasis (such as manifested as cerebral edema and/or progressive growth); Central nervous system conversion

Individuals limited to the brain and cerebellum can participate in screening if they meet the following conditions:

a. Asymptomatic brain metastases (asymptomatic central nervous system progressive symptoms caused by brain metastases, also not necessary) Using corticosteroids or antiepileptic drugs for treatment; b. Symptoms stabilize for at least 2 weeks after radiotherapy for brain metastases, and corticosteroids or antiepileptic drugs are discontinued Drug discontinuation for at least 2 weeks;

* Evidence of significant coagulation disorders or other significant bleeding risks:

  1. History of intracranial hemorrhage or spinal cord hemorrhage;
  2. Patients with tumor lesions invading large blood vessels and having a significant risk of bleeding;
  3. Within the 6 months prior to the start of the study treatment, there have been incidents of thrombosis or embolism (asymptomatic and none) Except for intramuscular venous thrombosis that requires treatment, there is no absorption during follow-up examination, or significant vascular disease is present (For aortic aneurysm, aortic dissection, etc. that require surgical repair);
  4. Clinically significant hemoptysis or tumor development for any reason within the first 3 months prior to starting the study treatment Blood;
  5. Within 14 days prior to the start of the study, use anticoagulant therapy for therapeutic purposes (with low prophylactic use) Excluding molecular weight heparin;
* Past or current active autoimmune diseases or immunodeficiency, including but not limited to severe muscle disease Weakness, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammation Sexually transmitted bowel disease, antiphospholipid antibody syndrome, Wegener's granulomatosis, Sj ö gren syndrome, Grimm Barr syndrome Li syndrome or multiple sclerosis; Except for: a Autoimmune related hypothyroidism Subjects with a history of withdrawal and currently taking thyroid replacement hormone; b. Stable status receiving insulin treatment 30% of subjects with type I diabetes.
* Lesions limited to subjects with eczema, psoriasis, chronic simple lichen, and vitiligo on the skin (if diseased)

When the damage has already affected parts or organs outside the skin (such as psoriasis, arthritis, etc.), it cannot be included in the group:

i. Fever of unknown origin>38.5 ℃ (fever caused by tumor can be included in the group);

* Within 6 months prior to starting the study of drug therapy, the following situations occurred:

  1. Suffering from congestive heart failure, severe/unstable angina, cerebrovascular accident, New York, USA Cardiac insufficiency classified by the Society of Cardiology (NYHA) as Grade II or above (including Grade II), Or other structural heart diseases that have been determined by researchers to be at high risk;
  2. History of abdominal fistula, tracheoesophageal fistula, gastrointestinal perforation, or abdominal abscess;
  3. There is uncontrollable tumor related pain, and if painkillers are needed, they should be stable during screening A prescribed pain relief treatment plan; Asymptomatic metastatic lesions, if further grown, may lead to Causing functional impairment or stubborn pain (such as epidural metastases that are currently unrelated to spinal cord compression), If appropriate, local treatment should be considered before screening;
* Within the 5 years prior to starting the research on drug therapy, if there were other active malignant tumors, local treatment may be necessary Except for malignant tumors that have been treated and cured (such as basal cell or squamous cell carcinoma of the skin, superficial or non malignant) Invasive bladder cancer cancer, cervical carcinoma in situ, breast intraductal carcinoma in situ, thyroid papillary carcinoma);
* Individuals who have received allogeneic hematopoietic stem cell transplantation or organ transplantation in the past;
* Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS);
* Syphilis antibody positive and active syphilis infection present;
* Individuals with active pulmonary tuberculosis or a history of pulmonary tuberculosis infection that cannot be controlled after treatment;
* 20 HBsAg or HBcAb positive, and HBV-DNA>2000 IU/mL (for For patients with HBV DNA>500 IU/mL, the subject must agree to at least 7 days prior to the start of the study drug Continuously receiving antiviral treatment other than interferon during the research period is necessary to participate in screening; HCV antibodies Positive and HCV-RNA higher than the lower limit of detection in the experimental center (if the center is unable to detect HCV) RNA, acceptable external hospital results, relevant reports should be provided);
* Expected to receive any other form of anti-tumor drug treatment during the trial period;
* Known to have a history of alcohol abuse, psychotropic substance abuse, or drug use;
* Individuals with mental disorders or poor compliance;
* Pregnant or lactating women
* According to the judgment of the researchers, the basic condition of the subjects may increase their risk of receiving study drug treatment,Or confusion caused by the occurrence of toxic reactions and the explanation of AE;
* Other researchers deemed it unsuitable to participate in this experiment;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival(PFS) | 5 years from first patient randomized
  The time from the start of randomization until the first occurrence of disease. progression or death from any cause, whichever occurs first.
overal survival time(OS) | 5 years from first patient randomized
  The time from randomization to death from any cause

SECONDARY OUTCOMES:
Adverse events | Duration of time from the start of treatment to the end of study, assessed up to 5 years
  The type, frequency, severity, and degree of treatment-related adverse events (according to CTCAE version 5.0)
objective response rate(ORR) | Duration of time from the start of treatment to the end of study, assessed up to 5 years
  The proportion of patients with a complete or partial response
Disease control rate(DCR) | Duration of time from the start of treatment to the end of study, assessed up to 5 years
  the proportion of patients with a complete response, partial response, or stable disease

IPD SHARING:
Plan to Share IPD: No